CLINICAL TRIAL: NCT00234546
Title: A 24-week Prospective, Multicentre, Randomised, Double-blind, Placebo Controlled Study of Dysport® Injection for the Treatment of Upper Limb Spasticity in Early Stroke.
Brief Title: Asian Botulinum Clinical Trial Designed for Early Stroke Spasticity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-38-52120-713
Record Dates: First submitted 2005-10-06; First posted 2005-10-07 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Muscle Spasticity; Cerebrovascular Accident
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Dysport
  Interventions: Biological: Botulinum toxin type A
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — 1 injection, 500 U at day 0. The study will last for 6 months in each patient.
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: 1
Drug: Placebo — 1 injection at day 0. The study will last for 6 months in each patient.
  Arms: 2

SUMMARY:
The aim of this clinical study is to investigate the efficacy and safety of Dysport® in patients with early onset of upper limb spasticity within 2-12 weeks after stroke.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke according to the World Health Organisation criteria (previous transient ischaemic attack or clinically silent infarct on CT/MRI is not counted as previous stroke)
* CT/MRI scan required to classify ischaemic / haemorrhagic stroke
* Patient recruited 2-12 weeks after stroke
* Modified Ashworth Spasticity Score 1+ or above in either elbow or wrist joint

Exclusion Criteria:

* The patient has bleeding disturbances or having used coumarin derivatives
* The patient is currently receiving drugs affecting neuromuscular transmission
* Co-existing severe systemic illness which may adversely affect the functional outcome
* Pre-existing neuromuscular junction disease or any neurogenic disorders which can interfere with spasticity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2003-02; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Reduction of spasticity assessed by changes of the Modified Ashworth Spasticity Score from baseline of elbow and wrist flexors in supine anatomical position | week 4

SECONDARY OUTCOMES:
Improvement of neurologic outcome (mobility and function), evaluated by Modified Ashworth Scale, Barthel Index, Modified Rankin scale, Functional scale (Motor Assessment Scale) | weeks 4, 8, 12 & 24
Voluntary and passive joint range of motion goniometer assessment | weeks 4, 8, 12 & 24
Pain Assessment using visual analogue scale for pain | weeks 4, 8, 12 & 24

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (5):
- Prince of Wales Hospital, Shatin, Hong Kong
- University Hospital of Malaya Medical Centre, Kuala Lumpur, Malaysia
- University of Santo Tomas, Manila, Philippines
- TTSH Rehabilitation Centre, Singapore, Singapore
- Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Result] Rosales RL, Kong KH, Goh KJ, Kumthornthip W, Mok VC, Delgado-De Los Santos MM, Chua KS, Abdullah SJ, Zakine B, Maisonobe P, Magis A, Wong KS. Botulinum toxin injection for hypertonicity of the upper extremity within 12 weeks after stroke: a randomized controlled trial. Neurorehabil Neural Repair. 2012 Sep;26(7):812-21. doi: 10.1177/1545968311430824. Epub 2012 Feb 27. PMID 22371239